CLINICAL TRIAL: NCT02553668
Title: Proteomics for Identification of Hyperoxia-induced Changes in Protein Expression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Stefan Braunecker, Anesthesiologist, University Hospital of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-109
Record Dates: First submitted 2015-07-09; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Hyperoxia
Keywords: Proteomics; Oxygen; Pathways
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperoxia (Experimental): Participants receive 100% oxygen
  Interventions: Drug: Oxygen (FiO2 1,0); Device: Facemask

INTERVENTIONS:
Drug: Oxygen (FiO2 1,0) — Participants will inhale Oxygen (FiO2 1,0) via Facemask for 3 hours.
Device: Facemask

SUMMARY:
Aim of the present study is to investigate the influence of hyperoxia on the protein expression using the differential analysis of protein expression in tissues (proteomics). In the study, blood and urine samples will be collected from participants who undergo a short term hyperoxia using 100% oxgen for 3 hours.

Here, gel electrophoresis, protein separation and mass spectroscopy allow to identify affected proteins. Based on these results, different induction factors of proteins will be determined and then assessed using a bioinformatic network analysis regarding the cellular influence.

DETAILED DESCRIPTION:
Oxygen is necessary to sustain human life and is used for energy production by oxidation in the mitochondria. Application of oxygen not only increases saturation in the patient's blood, but also has various secondary effects. It is therefore used to treat diseases that impairs body's ability to take up and use oxygen. But even healthy people can suffer from hypoxia when they ascend to high altitude. Here, altitude sickness can lead to potentially fatal complications such as high altitude cerebral edema or high altitude pulmonary edema. Since hypoxia can have disastrous consequences, hyperoxia is often tolerated in many pre- and in-hospital situations.

Whereas the effects of hypoxia are well studied, especially publications in the last decade have led to a new perspective on oxygen application. Besides pathophysiological changes as the peripheral vasoconstriction or reduction of contractility, especially changes on cellular level seem to be of great importance. Here, oxidative stress and change of protein synthesis in various organ are focus of current studies.

The differential analysis of protein expression in tissues (proteomics) is an important approach for better understanding of the negative effects of hyperoxia. Especially for patients with long-term high oxygen demand the knowledge of cellular changes during hyperoxia can result in new therapeutic approaches and a reduction in the rate of complications.

In the present molecular biology study urine and blood samples of healthy volunteers will be collected at specified times after short-term exposure to oxygen. These samples will be analyzed after the study using the differential analysis of protein expression. The aim of this study is to investigate the effects of oxygen on the cell functions by analyzing and subsequent bioinformatic processing of differentially regulated proteins in the blood and urine.

After checking the inclusion and exclusion criteria biometric data of the test persons are collected.

Before short-term hyperoxia a sample collection of blood and urine will be performed. Here the participants are taken 5 ml of venous blood from the cephalic vein under sterile conditions. To obtain the urine sample spontaneous urine of participants is used. The samples are immediately centrifuged and flash frozen at -80°C. In order to exclude impairment of the lung prior to the short-term hyperoxia a pulmonary function test is carried out by using a hand spirometer.

To induce hyperoxia subjects inhale 100% oxygen for 3 hours through a face mask.

After carrying out the short term hyperoxia the follow up phase takes place. In this phase blood and urine samples from the subjects will be obtained directly after the hyperoxia (T0), on day 1 (T1), day 3 (T3), day 7 (T7), day 14 (T14), day 21 (T21) and day 28 (T28) after oxygen exposure. All samples will be centrifuged immediately after collection and flash frozen at -80 ° C. To exclude hyperoxia-induced lung impairments, a spirometry is performed during the follow up.

After the samples of all subjects were collected the analysis of the samples will be carried out using Proteomics.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1
* >18 years
* < 50 years

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) > 1
* pregnant
* <18 years
* > 50 years
* frequent or recent drug intake

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of proteomics changes before and after short-term hyperoxia | 4 weeks

SECONDARY OUTCOMES:
Spirometry Results: Forced vital capacity (FVC) [L] | 2 days
  Spirometry will be used as a measure of safety to rule out adverse events of oxygen to the lung.
Spirometry Results: Forced expiratory volume at one second (FEV1) [L] | 2 days
  Spirometry will be used as a measure of safety to rule out adverse events of oxygen to the lung.
Spirometry Results: Forced expiratory flow (FEF25-75) [L/s] | 2 days
  Spirometry will be used as a measure of safety to rule out adverse events of oxygen to the lung.
Spirometry Results: Peak expiratory flow (PEF) [L/s] | 2 days
  Spirometry will be used as a measure of safety to rule out adverse events of oxygen to the lung.
Vital parameter: Respiratory rate (RR) [1/min] | 3 hours
  Vital parameters will be used as a measure of safety to rule out adverse events of oxygen to the vascular system.
Vital parameter: Heart rate (HR) [1/min] | 3 hours
  Vital parameters will be used as a measure of safety to rule out adverse events of oxygen to the vascular system.
Vital parameter: Blood pressure (BP) [mmHg] | 3 hours
  Vital parameters will be used as a measure of safety to rule out adverse events of oxygen to the vascular system.
Vital parameter: Oxygen saturation (SpO2) [%] | 3 hours
  Vital parameters will be used as a measure of safety to rule out adverse events of oxygen to the vascular system.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Braunecker, M.D., Principal Investigator — Universityhospital of Cologne

REFERENCES:
- [Background] Spelten O, Wetsch WA, Wrettos G, Kalenka A, Hinkelbein J. Response of rat lung tissue to short-term hyperoxia: a proteomic approach. Mol Cell Biochem. 2013 Nov;383(1-2):231-42. doi: 10.1007/s11010-013-1771-y. Epub 2013 Aug 11. PMID 23934118
- [Background] Hinkelbein J, Feldmann RE Jr, Kalenka A. Time-dependent alterations of cerebral proteins following short-term normobaric hyperoxia. Mol Cell Biochem. 2010 Jun;339(1-2):9-21. doi: 10.1007/s11010-009-0365-1. Epub 2010 Jan 5. PMID 20049628